CLINICAL TRIAL: NCT00636649
Title: Escitalopram Treatment of Night Eating Syndrome: a Randomized Controlled Trial
Brief Title: Escitalopram Treatment of Night Eating Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: St. Louis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00007133; LXP-MD-128A
Record Dates: First submitted 2008-02-03; First posted 2008-03-14 (Estimated); Results first posted 2013-05-06 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-05

CONDITIONS: Night Eating Syndrome
Keywords: Eating disorder
MeSH Terms: conditions — Night Eating Syndrome; Feeding and Eating Disorders | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Escitalopram
  Interventions: Drug: Escitalopram
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — 10-20 mg
  Arms: A
Drug: Placebo — Placebo
  Arms: B

SUMMARY:
Night-Eating Syndrome (NES) is an eating disorder characterised by excessive eating at night, sleep disturbance and morning anorexia. This 12-week study examines the effect of escitalopram on symptoms of NES.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Presence of NES
* BMI 25-50

Exclusion Criteria:

* History of schizophrenia or other psychoses
* History of bipolar disorder, anorexia nervosa, bulimia, binge eating disorder
* Current major depressive disorder
* Suicidal ideation
* Psychotropic drugs in the past month
* Drugs or herbal remedies that significantly affect body weight, current participation in a weight loss program, currently following a specialized diet (e.g., Atkins, Zone, etc)
* Lack of benefit with SSRI treatment for NES
* Serious or unstable medical illness
* Allergy or hypersensitivity to escitalopram
* Pregnant, breast-feeding, or planning pregnancy in the next six months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10; Primary Completion 2010-08 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kishore Gadde, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Saint Louis University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Vander Wal JS, Gang CH, Griffing GT, Gadde KM. Escitalopram for treatment of night eating syndrome: a 12-week, randomized, placebo-controlled trial. J Clin Psychopharmacol. 2012 Jun;32(3):341-5. doi: 10.1097/JCP.0b013e318254239b. PMID 22544016

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at Duke University Medical Center and Saint Louis University between 2008 and 2010.
Groups:
- Escitalopram: Escitalopram was started at 10 mg/d and the dose was increased to 20 mg/d after 4 weeks.
- Placebo: Dosing of matching placebo was identical.
Period: Overall Study
Arm/Group | Escitalopram | Placebo
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (13.7) | 44.8 (12.3) | 45.0 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Night Eating Questionnaire
Description: The Night Eating Questionnaire (NEQ) is a 14-item self-report scale designed to assess the symptoms of NES including nocturnal ingestions, evening hyperphagia, morning anorexia, and mood/sleep. Scores range from 0-56, with higher scores indicative of greater severity. The NEQ has an acceptable internal consistency reliability (.70). A cut-score of 25 has been shown to yield a positive predictive value of .62.
Time Frame: baseline, 12 weeks
Population: Data were analyzed as intent-to-treat with all 40 patients included in the analysis. Primary endpoint was change in the NEQ total score, i.e., difference between values between Week 12 (study exit) and baseline. Analysis of covariance was the primary statistical procedure with baseline NEQ score and baseline BMI as covariates.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -13.0 (1.6) | -10.6 (2.2)

2. Secondary Outcome: Change in Beck Depression Inventory II (BDI-II) Score
Description: The BDI-II is a 21-item self-report questionnaire designed to measure cognitive, somatic, and behavioral aspects of depression. Scores range from 0 to 63, with higher scores indicating a higher level of depressive symptoms.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -2.4 (1.2) | -3.5 (1.5)

3. Secondary Outcome: Change in Coping Inventory for Stressful Situations (CISS)
Description: TASK = task-oriented coping; EMOT = emotion-oriented coping; AVD = avoidance-focused coping; Avoidance-focused coping may be divided into two subtypes: DIS = distraction-oriented coping; SOC = social diversion-oriented coping. CISS is a 48 item self-report measure used to measure responses to stressful situations rated for frequency on a 5 point Likert scales ranging from1, not at all to 5, very much. This measure assesses three coping styles: Task-Oriented, Emotion-Oriented, and two types of Avoidance-Oriented coping (Social Diversion and Distraction). There are 16 items on each of the primary scales (task, emotion, avoidance) and 5 on social diversion and 8 on distraction. Scores are summed for each subscale and then converted to gender-corrected t-scores with a mean of 50 and a standard deviation of 10. T-scores on the CISS range from a low of 25 (1st percentile) to 75 (99th percentile). Higher scores indicate more adaptive levels of coping.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: t-scores
Arm/Group | Placebo | Escitalopram
Number analyzed (Participants) | 20 | 20
t-scores
  CISS-TASK | 2.35 (3.50) | 1.75 (1.37)
  CISS-EMOT | 1.25 (2.82) | -1.45 (1.37)
  CISS-AVD | 0 (3.31) | 2.60 (1.10)
  CISS-DIS | 3.40 (2.42) | 1.95 (1.33)
  CISS-SOC | -2.45 (2.08) | 2.15 (1.62)
Statistical Analysis 1: Comparison: Placebo vs Escitalopram; CISS-TASK; Test type: Superiority or Other; p = 0.993, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Escitalopram; CISS-EMOT; Test type: Superiority or Other; p = 0.185, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Escitalopram; CISS-DIS; Test type: Superiority or Other; p = 0.196, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Escitalopram; CISS-AVD; Test type: Superiority or Other; p = 0.759, ANCOVA
Statistical Analysis 5: Comparison: Placebo vs Escitalopram; CISS-SOC; Test type: Superiority or Other; p = 0.396, ANCOVA

4. Secondary Outcome: Change in Perceived Stress Scale (PSS)
Description: The Perceived Stress Scale (PSS) measures the overall level of stress. This instrument contains 14 items accessing overall appraisals of stress in the past month. Minimum score (best value)=0. Maximum score (worst value)=56. A higher score indicates greater stress.
Time Frame: 12 weeks
Population: Participants who completed PSS assessment at baseline and week 12.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Escitalopram
Number analyzed (Participants) | 20 | 18
units on a scale | -0.55 (1.42) | -2.11 (1.39)
Statistical Analysis 1: Comparison: Placebo vs Escitalopram; Test type: Superiority or Other; p = 0.579, ANCOVA

5. Secondary Outcome: Change in Three Factor Eating Questionnaire (TFEQ)
Description: The TFEQ (also known as the Eating Inventory) measures dimensions of eating behavior including cognitive restraint of eating, disinhibition, and hunger using a combination of dichotomous questions, 4-point likert scales, and one 5-point likert scale. Restraint is comprised of the responses to 21 questions with possible scores ranging from 0 to 21 (Low scores for all scales indicate an uninhibited eating behavior.). Disinhibition is comprised of the responses to 16 questions with possible scores ranging from 0 to 16 (High scores indicate an uninhibited eating behavior strongly depending on external cues). Hunger is comprised of the responses to 14 questions with possible scores ranging from 0 to 14 ( Low scores indicate an eating behavior strongly depending on feelings of hunger.).
  RES = Restraint Subscale; DIS = Disinhibition Subscale; HUN = Hunger Subscale
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Escitalopram
Number analyzed (Participants) | 20 | 20
units on a scale
  TFEQ-RES | 2.95 (1.12) | 1.85 (0.56)
  TFEQ-DIS | -0.85 (0.73) | -1.50 (0.61)
  TFEQ-HUN | -1.60 (0.76) | -1.75 (0.63)
Statistical Analysis 1: Comparison: Placebo vs Escitalopram; TFEQ-RES; Test type: Superiority or Other; p = 0.225, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Escitalopram; TFEQ-DIS; Test type: Superiority or Other; p = 0.498, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Escitalopram; TFEQ-HUN; Test type: Superiority or Other; p = 0.724, ANCOVA

6. Secondary Outcome: Number of Participants With a Clinical Global Impression - Improvement (CGI-I) Score ≤ 2
Description: The CGI-I scale is a clinician rating of overall therapeutic effect ranging from 1 (very much improved) to 7 (very much worse) since commencing treatment.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 20 | 20
participants | 12 | 7

7. Secondary Outcome: Change in Lipid Panel
Time Frame: Baseline,12 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 20 | 20
mg/dL
  HDL | -2.8 (1.8) | -2.2 (1.8)
  LDL | -3.9 (4.4) | 2.8 (4.5)
  Triglycerides | 27.5 (26.3) | -14.0 (15.6)
  total cholesterol | -4.5 (5.2) | -2.3 (4.5)

8. Secondary Outcome: Change in Beck Anxiety Inventory (BAI) Score
Description: The Beck Anxiety Inventory (BAI) is a 21-item self-report measure of anxiety. Scores range from 0 to 63, with higher scores indicative of higher levels of anxiety.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -1.5 (0.8) | -1.8 (0.9)

9. Secondary Outcome: Change in Glucose
Time Frame: Baseline, 12 Week
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 20 | 20
mg/dL | 3.9 (6.3) | 7.6 (4.6)

10. Secondary Outcome: Change in Weight
Time Frame: Baseline, 12 week
Measure: Mean (Standard Error); unit: kg
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 20 | 20
kg | -0.43 (0.7) | 1.12 (0.6)

11. Secondary Outcome: Number of Participants Who no Longer Meet the NESHI Criteria
Description: The Night Eating Syndrome History and Inventory (NESHI) is an unpublished, semistructured interview used to confirm a diagnosis of NES. It assesses a typical 24-hour food intake, including a recall of all meals and snacks, and sleeping patterns. Based on the recall of all meals and snacks, the interviewer judged whether ≥25% of the daily caloric intake was eaten after the evening meal and how often nocturnal ingestions occurred. The NEQ items were reviewed and informed by the dietary recall during the interview, and a new total score was tallied. A final score of ≥25 for the NEQ items, as reviewed during the NESHI, was used as the criterion for NES.
Time Frame: Week 12
Measure: Number; unit: participants
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 20 | 20
participants | 16 | 12

12. Secondary Outcome: Number of Participants Who Had a 50% Reduction in NEQ Scores
Description: The Night Eating Questionnaire (NEQ) is a 14 item self-report scale designed to assess the symptoms of NES including nocturnal ingestions, evening hypcrphagia, morning anorexia, and mood/slccp. Scores range from 0 to 56, with higher scores indicative of greater severity.
Time Frame: Week 12
Measure: Number; unit: participants
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 20 | 20
participants | 7 | 6

ADVERSE EVENTS:
Arm/Group | Escitalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 9/20 | 7/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=20) | Placebo (N=20)
headache (Nervous system disorders) | 5 | 2
drowsiness (Psychiatric disorders) | 4 | 0
gastrointestinal symptoms (Gastrointestinal disorders) | 0 | 2
upper respiratory infection / seasonal allergies (Immune system disorders) | 3 | 3
fatigue (General disorders) | 3 | 0
Sexual Dysfunction (Reproductive system and breast disorders) | 2 | 0
cognitive symptoms (Nervous system disorders) | 2 | 0 — difficulty concentrating, feeling spacey

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No